CLINICAL TRIAL: NCT02198508
Title: The Shuttle Effect : Combination Therapy With Deferiprone and Deferasirox in Transfusion-dependent Thalassemia Patients.
Brief Title: Clinical Trial of Deferasirox Combination Treatment With Deferiprone In Thalassaemia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Ching-Tien Peng, superintendent, China Medical University, Taiwan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DMR-096-IRB-037
Record Dates: First submitted 2014-07-19; First posted 2014-07-23 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Beta-thalassemia Major
MeSH Terms: conditions — beta-Thalassemia | interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DFX single treatment (Active Comparator): a single oral dose of DFX 30 mg/kg once daily, (Exjade®, Novartis Pharmaceuticals Corporation, USA )
  Interventions: Drug: DFX(Deferasirox)
- DFP single treatment (Active Comparator): single oral dose of DFP 40 mg/kg/day twice a day, (Kelfer®, Cipla Ltd., India)
  Interventions: Drug: DFP(Deferiprone)
- combination treatment (Experimental): sequential oral doses of DFX 30 mg/kg/d, DFP 40 mg/kg/d and DFP 40 mg/kg/d (dosing interval: seven hours).
  Interventions: Drug: DFX(Deferasirox); Drug: DFP(Deferiprone)

INTERVENTIONS:
Drug: DFX(Deferasirox)
  Other Names: Exjade®, Novartis Pharmaceuticals Corporation, USA
  Arms: DFX single treatment; combination treatment
Drug: DFP(Deferiprone)
  Other Names: Kelfer®, Cipla Ltd., India
  Arms: DFP single treatment; combination treatment

SUMMARY:
Background: Three iron chelators now available on the market differ in toxicity and organ specificity; evidence on standardized chelation protocol remains inconclusive, but patients with transfusion-dependent beta-thalassemia treated with DFO infusion show significant differences in the limitations of daily activities, physical activity, and quality of life when treated with oral chelator. With licensing of DFP in America, it is reasonable to combine DFP with DFX. Patients find two oral chelators more acceptable than one oral and one injectable. This pilot study rates use of DFP for improving iron excretion profile of deferasirox.

Methods: The investigators enrolled 13 beta-thalassemia patients in China Medical University Children's Hospital in May 2009-October 2011. Five refused to take part in pharmacokinetics; they only participated in iron excretion study. Seven with irregular bowel function were unable to collect feces in the screening period as baseline data. Subjects were randomly assigned and rotated to undergo all treatments (with informed consent): (A) single oral dose of DFX 30 mg/kg once daily, (B) single oral dose of DFP 40 mg/kg twice a day, (C) oral doses of DFX and DFP administered sequentially (DFX 30 mg/kg/d, deferiprone 40 mg/kg/d and deferiprone 40 mg/kg/d at 7-hour intervals). Three-day drug dosage was followed by four-day washout. Collections of urine and stool proceeded 24 hours per day, each analyzed separately. Through a venous catheter, serial blood samples (1 mL/each sampling) were collected in glass tubes containing heparin as anticoagulant at Time 0 (pre-dosing) and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 6, 7, 8, 10, 12 and 24 hours after dose; plasma concentrations of DFP and DFX were measured.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* serum ferritin greater than 2000 ng/mL,
* serum creatinine within normal range for a measuring laboratory
* platelet count exceeding 140000/mm3
* body weight at least 40 Kg
* None had a history of clinical significant of gastrointestinal, hepatic, renal, endocrine, oncologic, infectious, pulmonary or cardiovascular disease

Exclusion Criteria:

* HIV positive, history of immunologic hypersensitivity to any medication
* women pregnant or breast feeding
* drug or alcohol abuse
* patients showed abnormal or irregular bowel function (defined as more than three bowel movements a day or less than one bowel movement every other day)
* receiving warfarin, digoxin, or anti-arrhythmic or antiseizure medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-07; Primary Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
iron excretion from urine and feces by flame atomic absorption spectroscopy | 25-days
  Collections of urine and stool (made 24 hours a day) were analyzed separately.

SECONDARY OUTCOMES:
drug concentration in plasma by pharmacokinetics analysis | 25-day
  Through a venous catheter, serial blood samples (1 mL/each sampling) were collected into glass tubes containing heparin as an anticoagulant at time 0 (pre-dosing) and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 6, 7, 8, 10, 12 and 24 hours after dosing. Blood samples were centrifuged, with plasma collected and frozen at -20°C until analysis.